CLINICAL TRIAL: NCT00024570
Title: Interstitial Infusion of IL13-PE38QQR Cytotoxin in Recurrent Malignant Glioma: Phase I/II Study
Brief Title: Interstitial Infusion of IL13-PE38QQR Cytotoxin in Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IL13PEI-001; NCI-NABTT-9903; JHU-NABTT-9903
Record Dates: First submitted 2001-09-20; First posted 2001-09-21 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Malignant Glioma; Glioblastoma Multiforme; Anaplastic Astrocytoma; Mixed Oligoastrocytoma
Keywords: neurosurgery, craniotomy; convection-enhanced delivery; CNS interstitial infusion; recombinant toxins; malignant glioma, recurrent; catheter, stereotaxic; intratumoral therapy; positive pressure microinfusion
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma; Recurrence | interventions — IL13-PE38; Surgical Procedures, Operative

INTERVENTIONS:
Drug: IL13-PE38QQR
Procedure: targeted fusion protein therapy
Procedure: surgery

SUMMARY:
IL13-PE38QQR is an oncology drug product consisting of IL13 (interleukin-13) and PE38QQR (a bacteria toxin). IL3-PE38QQR is a protein that exhibits cell killing activity against a variety of IL13 receptor-positive tumor cell lines indicating that it may show a therapeutic benefit. In reciprocal competition experiments, the interaction between IL13-PE38QQR and the IL13 receptors was shown to be highly specific for human glioma cells.

IL13-PE38QQR will be infused in two courses of 96 hours each, eight weeks apart, directly into the malignant brain tumors of patients to determine the dose of drug these patients can tolerate. After that, the selected dose will be studied to give an estimate of the response rate, response duration, time to response, and survival after infusing that dose of IL13-PE38QQR into the recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the toxicities and maximum tolerated dose of IL13-PE38QQR delivered by continuous infusion into malignant glioma over 96 hours, in two courses eight weeks apart.

II. Estimate the response rate, response duration, time to response, and survival after interstitial infusion of IL13-PE38QQR into recurrent malignant glioma.

III. Describe the toxicities of interstitial infusion of IL13-PE38QQR at the selected dose.

PROTOCOL OUTLINE: Patients are expected to receive two IL13-PE38QQR infusions at 8-week intervals. For each course, drug will be infused through each of two catheters; infusion rate will be held constant during a 96-hour infusion.

In Phase I, the dose of IL13-PE38QQR will be increased by increasing the IL13-PE38QQR concentration in stepwise fashion, while holding infusion volume and duration constant. Three patients will be treated at each dose level until the maximum tolerated dose (MTD) is reached, and an additional three patients are treated at that level. In Phase II, patients will be treated at the selected MTD.

PROJECTED ACCRUAL: In Phase I, up to 30 patients will be treated. In Phase II, up to 35 patients will be treated.

ELIGIBILITY:
Disease Characteristics

* Must have had surgery (or biopsy) of a supratentorial brain tumor with pathologic diagnosis of malignant (grade 3 or 4) glioma, including anaplastic astrocytoma, glioblastoma multiforme and malignant mixed oligoastrocytoma. (Note: If diagnosis is dependent upon the Day 0 biopsy, pathology must be confirmed prior to start of IL13PE-38QQR infusion).
* Must have received cranial radiotherapy, with tumor dose of at least 48 Gy, completed at least 12 weeks prior to study entry.
* Must have radiographic evidence of recurrent or progressive supratentorial tumor compared with a previous study. The baseline tumor measurements must be determined within 2 weeks prior to study entry. The tumor must have a solid portion at least 1.0 cm but not more than 5.0 cm in maximum diameter. A maximum of one satellite lesion is permitted, if separated by less than 3 cm from the primary mass.
* Stereotaxic biopsy at study entry must confirm the presence of glioma.

Patient Characteristics

* Age 18 or greater.
* Karnofsky Performance Score must be at least 60.
* Hematologic status: Absolute neutrophils at least 1,500/mm^3; Hemoglobin at least 10 gm/dL; Platelets at least 100,000/mm^3; PT & PTT less than or equal to the upper limit of normal.
* Hepatic Status: Transaminases not more than 2.5 x upper limit of normal; Total Bilirubin not more than 2.0 mg/dL.
* Must have recovered from toxicity of prior therapy; at least 6 weeks elapsed since receiving nitrosourea-containing chemotherapy and 3 weeks since receiving any other chemotherapy.
* Must practice an effective method of birth control during the study.
* Must understand the investigational nature of this study and its potential risks and benefits, and must sign informed consent.
* No patients with more than two foci of tumor, tumor crossing the midline, or leptomeningeal tumor dissemination.
* No patients with impending herniation, spinal cord compression, or uncontrolled seizures.
* No patients who have received any localized antitumor therapy for the malignant glioma, either intralesional chemotherapy or focal radiotherapy (i.e. any form of stereotaxic RT or brachytherapy).
* No patients who are receiving concurrent chemotherapy or another investigational agent.
* No patients with prior or concurrent malignancy. (Patients with curatively treated carcinoma-in-situ or basal cell skin carcinoma OR who have been free of disease for at least 5 years are eligible).
* Female patients must not be pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2000-11; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Weingart, MD, Study Chair — The Johns Hopkins University
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - The Johns Hopkins University, Baltimore, Maryland
  - Henry Ford Health Systems, Detroit, Michigan
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania